CLINICAL TRIAL: NCT06302517
Title: Bispectral Index Monitoring Effect on Delirium Occurrence and Nursing Quality Improvement in Post-anesthesia Care Unit Patients Recovering From General Anesthesia
Brief Title: Bis Monitoring Effect on Delirium Occurrence and Nursing Quality Improvement Recovering From General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: K2020097
Record Dates: First submitted 2024-02-20; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Delirium, Postoperative
Keywords: bispectral index; postoperative delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-BIS-guided group (group C) (No Intervention): The depth of anesthesia was not monitored in the non-BIS-guided group (group C).
- BIS-guided group (group B) (Experimental): The BIS-guided group (group B) underwent intraoperative monitoring of BIS anesthesia depth
  Interventions: Device: BIS-guided

INTERVENTIONS:
Device: BIS-guided — underwent intraoperative monitoring of BIS anesthesia depth
  Arms: BIS-guided group (group B)

SUMMARY:
①Effects of BIS Index (BIS) monitoring on delirium incidence in Post-anesthesia care unit (PACU) in patients undergoing general anesthesia

②Effects of BIS BIS Index (BIS) monitoring on the quality of nursing care in the Post-anesthesia care unit (PACU)

DETAILED DESCRIPTION:
The effect of intraoperative anesthesia depth monitoring on delirium occurrence and improvement of nursing quality in the post-anesthesia care unit (PACU) remains unclear. We aimed to explore the effect of intraoperative anesthesia bispectral index (BIS) monitoring on delirium occurrence and improvement of nursing quality in the PACU for patients recovering from general anesthesia.

This randomized controlled trial included 120 patients, aged 20-80 years and classified as grades I-III according to the American Society of Anesthesiologists. The BIS-guided group (group B) underwent intraoperative monitoring of BIS anesthesia depth (maintained within the anesthetic range [40-60]). The depth of anesthesia was not monitored in the non-BIS-guided group (group C). The patients' vital signs were recorded at the beginning of the operation (T0), upon entering the PACU (T1), 15 min after extubation (T2), and after leaving the PACU (T3). Delirium score, emergence period (extubation and PACU observation times), and adverse events in the PACU were monitored. The nursing activity score (NAS) was used to evaluate the quality of care.

ELIGIBILITY:
Inclusion Criteria:

1. age ranging from 20 to 80 years
2. estimated operation time of 2 to 3 h
3. body mass index ≤30 kg/m2
4. normal preoperative heart, liver, lung, and renal function.

Exclusion Criteria:

1. Past cognitive impairment (dementia, cognitive impairment, mental illness or mental disorder)
2. Complex injuries: multiple fractures, chest and abdomen, pelvic and sacral trauma, head trauma, etc
3. Contraindications to intraspinal puncture (coagulation dysfunction, thrombocytopenia, intraspinal space occupation, puncture site infection, etc.)
4. Have a history of acute myocardial infarction or stroke within 3 months
5. Patients with severe liver dysfunction (Child-Pugh C) or renal failure
6. Contraindications to ketamine, such as malignant hypertension

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Ricker sedation-agitation scale | ￭evaluate immediately after recovery and tracheal intubation removal ￭every five minutes after that ￭take the highest value until the patient leave PACU
  Delirium was assessed using the Ricker sedation-agitation scale (SAS; unable to awaken = 1, very calm = 2, calm = 3, quiet cooperation = 4, agitated = 5, very agitated = 6, and dangerously agitated = 7)
The nursing activity score (NAS) | ￭at the begin of the patient enter PACU ￭end with the transfer out of the PACU ￭any nursing activitise will be scored
  The nursing activity score (NAS), consists of 23 nursing items in five aspects, including monitoring health care, supporting patients and their families, and managing nursing administration. Each item was assigned a score of 1.2-32.0 according to the percentage of time spent on the task during a nurse's working day. The higher the score, the greater the workload. The NAS score of each patient ranged from 0-177, and the assessment was conducted at the beginning of resuscitation in the PACU by a trained investigator according to the nursing work items on the NAS scale.
  According to the nursing records of patients, the nursing workload of PACU was evaluated and by the contents of NAS scale.
vital signs （Mean arterial pressure, heart rate, pulse oxygen saturation ） | ￭ at the beginning of surgery (T0), ￭at the time of extubation (T1), ￭10 minutes after extubation (T2), ￭at the time of leaving the PACU (T3: when patients were transferred from the PACU to the ward).
  collected from monitors （Mean arterial pressure, heart rate, pulse oxygen saturation）
Comparison of complications during the PACU period | The patients were transferred to PACU after surgery, the period during the PACU
  including postoperative delirium, nausea, vomiting, respiratory complications (e.g., SPO2 < 90%, arterial oxygen partial pressure < 60 mmHg, or interventions requiring mask compression, oxygen supply, manual mandibular ventilation, and intubation), cardiovascular-related complications (e.g., blood pressure exceeding 20% of preoperative value, HR < 120 beats /min or < 50 beats /min, emerging arrhythmia, and ischemia), severe pain, chills/hypothermia (skin temperature < 35 °C), and unplanned transfer to ICU.
The comprehensive satisfaction score | The patients were followed up 24 hours after surgery
  The comprehensive satisfaction score for anesthesia and nursing. The satisfaction score was categorized as excellent or generally poor based on criteria such as postoperative pain, influence on daily activities, and emotional stability. Excellent satisfaction indicated no or mild pain after surgery, no interference with daily activities, and emotional stability. General satisfaction indicated moderate pain that was tolerable, daily activities that were not affected or slightly reduced, and emotional stability. Poor satisfaction indicated moderate pain, significantly limited patient activities, low mood, or irritability.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital, School of Medicine, Zhejiang University, Jinhua, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No